CLINICAL TRIAL: NCT04364711
Title: Multi-centre EuRopean Study of MAjor Infectious Disease Syndromes (MERMAIDS) - Acute Respiratory Infections (MERMAIDS ARI) 2.0
Brief Title: EuRopean Study of MAjor Infectious Disease Syndromes Related to COVID-19
Acronym: MERMAIDS 2
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, MJM Bonten, Professor Medical Microbiology, UMC Utrecht
Other Study IDs: ReCoVer - MERMAIDS 2.0
Record Dates: First submitted 2020-04-20; First posted 2020-04-28 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; SARS-CoV 2
Keywords: acute respiratory infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background Rapid European COVID-19 Emergency Research response (RECoVER), is a project involving 10 international partners that has been selected for funding by the European Union under the Horizon 2020 research framework responding to call topic SC1-PHE-CORONAVIRUS-2020: Advancing knowledge for the clinical and public health response to the SARS-CoV-2 epidemic. MERMAIDS 2.0 is the hospital care study within RECOVER.

Rationale Detailed patient-oriented studies are needed to determine the spectrum of SARS-CoV-2 disease and the combined influences of age, comorbidities and pathogen co-infections on the development of severe disease, together with virological and immunological profiles. This research is key to understanding the pathophysiology and epidemiology of this new disease, as well as to identifying potential targets for therapeutic or preventive interventions.

Objective To establish the prevalence, disease spectrum and severity, clinical features, risk factors, spread and outcomes of novel 2019 coronavirus infection (SARS-CoV-2) in Hospital Care.

Study design Prospective observational cohort study in selected European countries.

Study population

Children and adults with 1) acute respiratory illness (ARI) presenting to hospital care during the SARS-CoV-2 epidemic (including both COVID-19 and non-COVID-19 patients) and 2) patients with confirmed COVID-19 infection, but with atypical presentation (non-ARI) or with nosocomial acquisition. Sites can optionally participate in the following tiers:

Tier 1 (Clinical data and biological sampling) - Clinical samples and data will be collected on enrolment day and then at scheduled time points.

Tier 2 (Clinical data an extended biological sampling). - incl. PBMC collection

Optional add-on study In a subset of sites and patients, COVID-19 positive patients will be followed post-discharge for 6 months to study clinical recovery and long-term sequelae Main study parameters/endpoints: Prevalence of COVID-19 among patients with acute respiratory illness. COVID-19 disease spectrum and host and pathogen risk factors for severity. Long-term sequelae of COVID-19 requiring hospital care. Proportion hospital-acquired COVID-19 infections and characteristics of nosocomial transmission.

Study Duration Scheduled 2 years and based on COVID-19 dynamics.

Nature and extent of the burden associated with participation, benefit and group relatedness This study is observational in nature. There will be no direct benefit to research participants. The study may include biological sampling in addition to sampling required for medical management. The results of the tests done on these samples may not contribute to improving the participant's health. Minimal inconvenience and discomfort to the participant may arise from study visits and biological sampling.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical suspicion of a new episode of acute respiratory tract infection.
2. Patient is admitted to hospital
3. Primary reason for hospital admission is clinical suspicion of a new episode of ARI
4. Onset of the following symptoms within the last 7 days: i. Sudden onset of self-reported fever OR temperature of ≥ 38°C at presentation AND ii. At least one respiratory symptom (cough, sore throat, runny or congested nose, dyspnea) AND iii. At least one systemic symptom (headache, muscle ache, sweats or chills or tiredness)

OR

Laboratory confirmed SARS-CoV-2 infection at the time of eligibility check.

Exclusion Criteria:

1. Inability to obtain consent from patient or surrogate
2. Previous enrollment in current study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a descriptive study of the clinical syndrome caused by SARS-CoV-2. Patients will only be considered for enrolment if appropriate local infection control and prevention measures are in place and can be maintained. In hospital, potential participants will be identified through hospital workers upon presentation at recruiting sites. The clinical research infrastructures of COMBACTE CLIN-NET will be used for site selection for an efficient establishment of a clinical network with broad European coverage providing access to a large patient population across all age groups and differing healthcare environments.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Pneumonia Severity indexes | 2 years
Need for supplemental oxygen; non-invasive or invasive mechanical ventilation; extra-corporeal life support | 2 years
Hospital - and ICU/HCU length of stay | 2 years
In-hospital mortality | 2 years
Activities of daily life, quality of life, variations in home living status and employment status | 2 years
Proportion of SARS-CoV2 positive patients | 2 years

CONTACTS AND LOCATIONS:
Locations (11):
- Tartu University, Tartu, Estonia
- Attikon Hospital, Athens, Greece
- Brescia Hospital, Brescia, Italy
- UMC Utrecht, Utrecht, Netherlands
- Nat.Inst. For Inf. Dis. Prof. Dr. Matei Bals, Bucharest, Romania
- Clinical Center of Podgorica, Podgorica, Serbia and Montenegro
- Serbia (2):
  - Clinical Center of Serbia, Belgrade
  - Clinical Center of Kragujevac, Kraljevo
- Spain (3):
  - Hospital Germans Trias i Pujol, Barcelona
  - Regional Hospital de Malaga, Málaga
  - Hospital Virgen Macarena, Seville